CLINICAL TRIAL: NCT04429178
Title: Portal Vein Pulsatility Flow in Pregnancy - a Pilot Study
Brief Title: Portal Vein Pulsatility Flow in Pregnancy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00774; qu19Buddeberg
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
Keywords: portal vein pulsatility; physiologic volume overload
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- women in the 1st trimester of pregnancy.
  Interventions: Other: ultrasound
- women in the 2nd trimester of pregnancy.
  Interventions: Other: ultrasound
- women in the 3rd trimester of pregnancy.
  Interventions: Other: ultrasound
- non-pregnant women
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — portal vein pulsatility fraction (percent) measured with ultrasound

SUMMARY:
This study is to investigate if portal vein pulsatility fraction can be measured in pregnancy and if it increases during the course of pregnancy as would be expected by the physiologic increase in blood volume that happens during pregnancy. Portal vein pulsatility fraction is measured in non-pregnant controls and in women in the 1st, 2nd and 3rd trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* American Society of Anesthesiologists (ASA) Class I and II
* Singleton pregnancy during 1st, 2nd or 3rd trimester or healthy non-pregnant females of childbearing age as controls

Exclusion Criteria:

* Inability to give informed consent
* Multiple gestation
* Significant co-morbidities (e.g. cardiac abnormalities, cardiac dysfunction, arrhythmias, severe asthma, renal insufficiency)
* High risk pregnancies (e.g. pre-eclampsia, gestational hypertension, HELLP, gestational diabetes)
* Body-Mass-Index (BMI) < 18kg/m2 or >40kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women attending either the anaesthetic preassessment clinic or the obstetric ultrasound clinic at University Hospital Basel.
  Non-pregnant healthy females fulfilling the inclusion criteria will be recruited by published advertisement at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Portal vein pulsatility fraction (percent) | single time-point at baseline
  Portal vein pulsatility fraction (percent)

SECONDARY OUTCOMES:
Inferior vena cava diameter (mm) | single time-point at baseline
  Inferior vena cava diameter (mm)
Inferior vena cava collapsibility index (percent) | single time-point at baseline
  Inferior vena cava collapsibility index (percent)
Hepatic venous flow (cm/sec) | single time-point at baseline
  Hepatic venous flow (cm/sec)
Right atrial and ventricular dimensions (cm) | single time-point at baseline
  Right atrial and ventricular dimensions (cm)
Tricuspid Annular Plane Systolic Excursion (TAPSE) (mm) | single time-point at baseline
  Tricuspid Annular Plane Systolic Excursion (TAPSE) (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Bigna Buddeberg, Dr. med., Principal Investigator — Department of Anesthesiology, University Hospital Basel
Locations (1):
- Department of Anesthesiology, University Hospital Basel, Basel, Switzerland